CLINICAL TRIAL: NCT01783431
Title: A Feasibility and Safety Study of Vaccination With Poly-ICLC and Peptide-pulsed Dendritic Cells in Patients With Metastatic and/or Unresectable Melanoma
Brief Title: Study of Vaccination With Poly-ICLC and Peptide-pulsed Dendritic Cells
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to low accrual.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101838
Record Dates: First submitted 2013-01-25; First posted 2013-02-04 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — poly ICLC; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Leukapheresis and Poly-ICLC (Experimental): Screening tests will be conducted to determine whether or not subjects can participate in this study. If subjects are eligible and choose to participate, they will have a procedure called leukapheresis. The leukapheresis product that is collected from you will be taken to a special lab at MUSC where it will undergo a process that will grow additional dendritic cells under controlled conditions in the lab. These cells will be given together with Poly-ICLC therapy when you begin study treatment. Some days you will receive both Poly-ICLC and dendritic cells, but on other days you will receive the Poly-ICLC by itself. After study treatment, subjects may be asked to return to MUSC approximately every 3 months for the first 2 years, then every 6 months thereafter for follow up procedures.
  Interventions: Drug: Poly ICLC; Procedure: leukapheresis

INTERVENTIONS:
Drug: Poly ICLC — Poly-ICLC is considered an investigational drug and has not been approved by the Food and Drug Administration (FDA) for treatment of your disease. It is currently being tested in clinical trials for brain tumors, lymphoma, human immunodeficiency virus (HIV) and prostate cancer. It is thought that Poly-ICLC, when used with dendritic cells as a vaccine therapy, may work to help the immune system fight disease.
Procedure: leukapheresis — Leukapheresis is a process in which white blood cells are collected from the body. These cells will be given together with Poly-ICLC therapy when subjects begin study treatment.

SUMMARY:
This study is for subjects with a type of skin cancer called melanoma. The main purpose of this study is to examine the safety of the study drug (Poly-ICLC) in patients with your disease. The study team would like to know about any side effects a patient may have when given the study drug. Another goal of the study is to determine if combining dendritic cells and the study drug can be possibly used as a vaccine for your disease.

DETAILED DESCRIPTION:
Dendritic cells are cells that are present in your body's immune system that help your body fight disease. This is a vaccine trial, as your own cells will be extracted (removed), treated in a lab, then re-administered to your body with the study drug in hopes of creating an immune response to the disease. It is not guaranteed that your disease burden will be reduced by participating in this trial.TScreening tests will be conducted to determine whether or not subjects can participate in this study. If subjects are eligible and choose to participate, they will have a procedure called leukapheresis. The leukapheresis product that is collected from you will be taken to a special lab at MUSC where it will undergo a process that will grow additional dendritic cells under controlled conditions in the lab. These cells will be given together with Poly-ICLC therapy when you begin study treatment. Some days you will receive both Poly-ICLC and dendritic cells, but on other days you will receive the Poly-ICLC by itself. After study treatment, subjects may be asked to return to MUSC approximately every 3 months for the first 2 years, then every 6 months thereafter for follow up procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of melanoma that is metastatic and/or unresectable. If the histologic diagnosis is based on a metastatic site, the histology must be compatible with melanoma.
* Patients must be HLA-A2 positivity by serological testing.
* Patients must have measurable disease per RECIST 1.1
* Patients may have had prior cancer therapy. Patients do not need to demonstrate progression to be considered for this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Age ≥ 18 years.
* Patient must have an expected life expectancy greater than 3 months.
* Signed, written IRB-approved informed consent.
* Acceptable organ function:
* Bilirubin ≤ 3 times upper limit of normal (CTCAE Grade 2 baseline)
* AST (SGOT), ALT (SGPT) ≤ 3 x ULN (CTCAE Grade 1 baseline)
* Serum creatinine ≤1.5 XULN (CTCAE Grade 1 baseline)
* Acceptable hematologic status:
* Absolute neutrophil count ≥ 1000 cells/mm3,
* Platelet count ≥ 75,000 (plt/mm3), (CTCAE Grade 1 baseline)
* Hemoglobin ≥ 9 g/dL.
* Urinalysis with no clinically significant abnormalities.
* PT and PTT ≤ 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT.

Exclusion Criteria:

* Patients must not have any serious uncontrolled acute or chronic medical condition that would interfere with this treatment. Examples would include active acute or chronic infection requiring antibiotics, uncontrolled cardiovascular, endocrine, or infectious disease.
* Patients must not have significant ongoing cardiac problems, myocardial infarction within the last six months, uncontrolled hypertension, unstable angina, uncontrolled arrhythmia or congestive heart failure.
* Surgery less than or equal to 14 days prior to study registration
* Patients who have had prior radiation or chemotherapy in which the last treatment administration is less than or equal to 28 days prior to registration. Patients who have had prior treatment with ipilimumab or Interleukin-2 will be allowed as long as this 28 day wash-out period is followed.
* Patients who are breast feeding or have a positive pregnancy test (if female).
* Patients with active CNS lesions are excluded (i.e., those with radiographically unstable, symptomatic lesions). However, a patient treated with stereotactic therapy or surgery is eligible if the patient remains without evidence of disease progression in the brain and is stable for 1 month. Whole brain radiotherapy is not allowed, with the exception of patients who have had definitive resection or stereotactic therapy of all radiologically detectable parenchymal lesions.
* Patients must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol treatment.
* Due to the undetermined effect of this treatment regimen in patients with HIV-1 infection and the potential for serious interaction with anti-HIV medications, patients known to be infected with HIV are not eligible for this study.
* Due to the possibility of harm to a fetus or nursing infant from this treatment regimen, patients must not be pregnant or nursing. Women and men of reproductive potential must have agreed to use an effective contraceptive method.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  - safety of this treatment by evaluating the qualitative and quantitative toxicities in this group of patients through adverse event reporting

SECONDARY OUTCOMES:
Feasibility | 2 years
  - feasibility of generating dendritic cells and administering these cells as a vaccine to patients
Anti-tumor Response | 2 years
  anti-tumor response after vaccination, measured by changes in tumor burden and overall survival
Immunological Responses | 2 years
  - immunological responses after vaccination (antigen-specific T cell cytokine production, antigen-specific T cell frequencies by tetramer analysis, and DTH reactions)

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Shirai, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States